CLINICAL TRIAL: NCT00509275
Title: A Phase Ib, Randomized, Double Blind, Placebo Controlled Study to Investigate the Pharmacokinetics, Safety and Efficacy of 3 Different Doses of W0027 and Placebo Capsules in Subjects With Clinically and Mycologically Proven MTTP
Brief Title: A Study to Evaluate Efficacy and Safety of Three W0027 Regimens in the Treatment of Moccasin Type Tinea Pedis (MTTP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W0027-08
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): W0027
  Interventions: Drug: W0027
- 2 (Experimental): W0027
  Interventions: Drug: W0027
- 3 (Experimental): W0027
  Interventions: Drug: W0027
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: W0027 — capsule
  Arms: 1; 2; 3
Drug: Placebo — Placebo
  Arms: 4

SUMMARY:
In this phase Ib, multi-centre, randomized, double-blind, placebo-controlled parallel group study, 120 subjects with moccasin type tinea pedis (MTTP) will be enrolled at approximately 11 centres in the USA, Canada and Australia.

The primary objective of the study is to assess the patient response to three W0027 regimens in subjects with MTTP. Secondary objectives include assessment of the safety, tolerability and skin and nail pharmacokinetics to the three Albaconazole regimens.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-65 years, who have been diagnosed with moccasin type tinea pedis (by positive dermatophyte culture, positive potassium hydroxide/calcofluor white preparation, and a Total Signs and Symptoms Score of at least 4).
* Females of childbearing potential must use contraceptive methods .

Exclusion Criteria:

* Subjects who are receiving any CYP3A substrates with potential for QT prolongation;
* have used systemic antifungal drugs within 30 days of first dose; or topical antifungals within 2 weeks of first dose.
* Also excluded are those who have a clinically significant medical condition.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the subject response to three W0027 regimens in subjects with MTTP. | Week 8

SECONDARY OUTCOMES:
The secondary objectives of this study are: To assess the safety and tolerability of three W0027 regimens in subjects with MTTP; To assess skin and nail pharmacokinetics of three Albaconazole doses in subjects with MTTP. | Skin and Plasma samples Week 0 (Visit 2) through to Week 8 (Visit 9), Nail samples Week 0 (Visit 2) Week 4(Visit 7) and Week 8(Visit 9)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Spelman, MD, Principal Investigator — South East Dermatology, South East Dermatology, Carina QLD 4152, Australia; Michael Freeman, MD, Principal Investigator — The Skin Centre, Benowa QLD 4217, Australia; Peter Foley, MD, Principal Investigator — Skin and Cancer Foundation, Carlton VIC 3053 , Australia; Stephen Shumack, MD, Principal Investigator — St George Dermatology and Skin Cancer Centre, Kogarah NSW 2217, Australia; Warren Weightman, MD, Principal Investigator — Dermatology on Ward, North Adelaide SA 5006, Australia; Debra Breneman, MD, Principal Investigator — University Dermatology Consultants, Inc., Cincinnati, OH, 45219, US; Eduardo Tschen, MD, Principal Investigator — Albuquerque, NM 87106, US; Yves Poulin, MD, Principal Investigator — Centre de Dermatologie de Québec Métropolitain, Quebec, QC, G1V 4X7, Canada; David Gratton, MD, Principal Investigator — International Dermatology Research Inc., Montreal, QC, H3H 1V4, Canada; Wayne Gulliver Gulliver, MD, Principal Investigator — NewLab Clinical Research, St. John's, NF, A1B 3E1, Canada; Steven Grekin, MD, Principal Investigator — 13450 East 12 Mile Road, Warren, MI 48088, US; Joseph Fowler, MD, Principal Investigator — Dermatology Specialists, 501 South Second Street, Louisville, KY 40202, US
Locations (9):
- United States (4):
  - Dermatology Specialists, Louisville, Kentucky
  - Warren, Michigan
  - Albuquerque, New Mexico
  - University Dermatology Consultants, Inc., Cincinnati, Ohio
- Australia (5):
  - St George Dermatology and Skin Cancer Centre, Kogarah, New South Wales
  - The Skin Centre, Benowa, Queensland
  - South East Dermatology, Carina, Queensland
  - Dermatology on Ward, North Adelaide, South Australia
  - Skin and Cancer Foundation, Carlton, Victoria